CLINICAL TRIAL: NCT05316727
Title: Electronic Nicotine Delivery Devices and Potential Progression to Acute Lung Injury
Acronym: ENDALI
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alison Morris, Professor, University of Pittsburgh
Other Study IDs: STUDY20020151; 5R01HL140963-04 (NIH)
Record Dates: First submitted 2022-02-23; First posted 2022-04-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Acute Lung Injury; Pulmonary Injury; Electronic Cigarette Use; Electronic Cigarette Related Lung Injury
Keywords: electronic nicotine delivery device (ENDD)
MeSH Terms: conditions — Acute Lung Injury; Lung Injury; Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Stool, oral wash, sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaping: At least weekly vape use over the past 3 months of the subjects unspecified product
- Non vapers: No previous history of vape use and no current history of smoking tobacco for controls

SUMMARY:
This is an observational - data and specimen collection study. There have been increasing reports of vaping-induced lung injury, including severe lung injury and rare cases of death. The mechanism by which vaping contributes to lung injury in susceptible persons is unknown, as is impact on chronic lung disease. The investigators aim to identify individuals with chronic electronic nicotine delivery device (ENDD) exposure and matched controls within our ongoing cohort of HIV+ and HIV-uninfected individuals, collect PFT data, bank respiratory and stool samples and collect clinical data for studies of clinical risk, inflammation, biomarkers, and the microbiome in the identification and modification of risk of progression to lung injury or chronic pulmonary disease.

DETAILED DESCRIPTION:
Participants will be consented and undergo collection of data and specimens as listed below.

* Vaping use will be determined by history.
* No administration, dispensing or use of any vape product will take place as part of the study.

Experimental procedures:

Respiratory questionnaires and data review:

Detailed data regarding smoking history, illicit drug use, ART and other medications, and medical history are obtained using standardized questionnaires and medical record review. The Modified Medical Research Council Dyspnea scale (MMRC), the St. George's Questionnaire(SGQT), Pulmonary questionnaire (PQ) and a Vaping questionnaire will be administered. These are paper and pencil questionnaires that inquire about respiratory symptoms, quality of life, and other lung related issues. Laboratory data including CD4 cell counts and HIV viral levels are obtained from the medical record.

Blood Sample collection:

The subject will be asked to provide a blood sample by venipuncture of approximately 110mls (7.4 tablespoon) at this study visit. The purpose of this collection is to have blood processed for serum, plasma, and PBMCS, and a portion stored for RNA to be used for future use. A hemoglobin and carboxyhemoglobin will be done in order to calculate the DLCO. A CBC will be done to determine overall health and possible infections.

Saliva Collection: Participants will be asked to produce saliva and spit it into a sterile conical.

Stool collection: The investigator will ask participants to provide a stool sample. The subject will be instructed on how to collect a stool specimen at home. The investigator will give the subject instructions and a kit that will provide all the supplies needed to collect the stool and return it via mail at their convenience.

Lung function testing (PFT):

If a PFT was completed for a research study in the past month, that data will be used instead of repeating the test. The routine lung function endpoints of FVC, FEV1, FEV1/FVC, and FEF25-75% will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system before and after bronchodilator administration. The system is calibrated for body temperature and pressure of saturated gas and volumes, per American Thoracic Society (ATS) standards . DLco will be measured using the automated single-breath procedure of the integrated testing system, which conforms with ATS standards. All testing will be reviewed by a physician associated with this study. If any concerns or abnormal results are discovered during this testing, a member of the research team will notify the subject or the subject's primary care physician, who will assess the need to provide additional evaluation.

Pregnancy Test: A urine pregnancy test will be performed on all women of child bearing potential. Men, and women who are post menopausal for at least 1 year or have been surgically made sterile will not have a pregnancy test.

Collection of the vape product used by the subject. Declining participation in this collection does not mean the subject can't participate in the study.

The product will be sent to the investigators research labs for potential chemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 80
* Participant in a previous HLRC study, or a participant in the HIV PACT clinic or referred by a PACCM physician
* At least weekly vape use over the past 3 months
* OR No previous history of vape use and no current history of smoking tobacco for controls
* negative pregnancy test (for women of child barring capabilities)

Exclusion Criteria:

* pregnancy or breast-feeding (urine pregnancy done on all females of child bearing potential- - - males and females who are at least 1 year post menopausal or surgically sterile will not be tested)
* Contraindication to pulmonary function testing (i.e. abdominal or cataract surgery within 3 months, recent myocardial infarction, etc.).
* Increasing respiratory symptoms or febrile (temperature >100.40F [380C]) within 4 weeks of study entry.
* Acute cardiopulmonary issue in the past 4 months.
* Uncontrolled hypertension at screening visit (systolic > 180 mm Hg or diastolic > 100 mm Hg) from an average of two or more readings. Subject may return for screening after blood pressure is controlled.
* Active cancer requiring systemic chemotherapy or radiation.
* Active infection of lungs, brain, or abdomen.
* Intravenous drug use or alcohol use that will impair ability to complete study investigations in the opinion of the investigator.
* subjects with an upper or lower respiratory tract infection
* Persons who have tested positive for Covid 19 in the past 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will leverage resources from an ongoing cohort of people living with HIV (PLWH) and HIV-uninfected community dwelling individuals as well as a growing dataset of individuals hospitalized with EVALI.
  individuals, males or females in all races, ethnicities, and socioeconomic backgrounds greater than 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Difference in pulmonary function comparing vaping and non vaping participants (1) | Before bronchodilation
  The routine lung function endpoints of FVC, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (2) | Before bronchodilation
  The routine lung function endpoints of FEV1, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (3) | Before bronchodilation
  The routine lung function endpoints of FEV1/FVC, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (4) | Before bronchodilation
  The routine lung function endpoints of FEF25-75%, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (PB1) | within 10 minutes after bronchodilation
  The routine lung function endpoints of FVC, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (PB2) | within 10 minutes after bronchodilation
  The routine lung function endpoints of FEV1 will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (PB3) | within 10 minutes after bronchodilation
  The routine lung function endpoints of FEV1/FVC, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in pulmonary function comparing vaping and non vaping participants (PB4) | within 10 minutes after bronchodilation
  The routine lung function endpoints of FEF25-75%, will be measured with the flow-volume loop recorder on a NDD Easy One Pro testing system.
Difference in diffusion capacity comparing vaping and non vaping participants | within 15 minutes after bronchodilation
  The routine lung function diffusion lung capacity for carbon monoxide (DLCO) will be measured.

SECONDARY OUTCOMES:
Change in inflammation | collected at one visit -will complete analysis in 2 years.
  The investigators will determine inflammation in sputum peripheral cytokine responses
Measurement of the inflammone in vaping and non vaping persons | collection at one visit - will complete analysis in 2 years.
  The investigators will use this cohort to evaluate biomarkers (type to be determined) of inflammation to determine if the investigator can identify specific HIV vapors phenotypes using novel decision tree analyses. The investigator will examine relationship of the inflammatory signature associated with vaping
comparison of microbial communities in stool | one stool collection at the subjects convenience - will complete analysis in 2 years.
  The investigators will use stool collected to compare bacterial function between vapers and non vapers

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh department of medicine division of Pulmonary, Allergy and Critical Care medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No